CLINICAL TRIAL: NCT01063036
Title: A Study of the Safety and Efficacy of Entecavir Plus Tenofovir in Adults With Chronic Hepatitis B Virus Infection With Previous Nucleoside/Nucleotide Treatment Failure
Brief Title: Efficacy and Safety Study of Entecavir Plus Tenofovir in Patients With Chronic Hepatitis B Who Failed Previous Treatment
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AI463-203; 2009-015705-40 (EudraCT Number)
Record Dates: First submitted 2010-02-03; First posted 2010-02-05 (Estimated); Results first posted 2014-02-13 (Estimated); Last update posted 2014-12-15 (Estimated); Status verified 2014-11

CONDITIONS: Chronic Hepatitis B
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — entecavir; Tenofovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Entecavir + Tenofovir (Experimental)
  Interventions: Drug: Entecavir; Drug: Tenofovir

INTERVENTIONS:
Drug: Entecavir — Tablets, Oral, 1 mg, once daily, 96 weeks
  Other Names: Baraclude®; BMS-200475
Drug: Tenofovir — Tablets, Oral, 300 mg, once daily, 96 weeks
  Other Names: Viread®

SUMMARY:
The purpose of this study is to show that the combination of entecavir and tenofovir, is effective and well tolerated in chronic hepatitis B patients who have failed previous treatment.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with chronic hepatitis B virus (HBV) infection; either hepatitis B-e antigen(HBeAg)-negative or HBeAg-positive
* Subjects must have a treatment failure to their current nucleoside/ nucleotide treatment regimen
* Prior entecavir and/or tenofovir monotherapy is allowed
* Subjects must have compensated liver function

Exclusion Criteria:

* Women who are pregnant or breastfeeding
* Evidence of decompensated cirrhosis
* Co-infection with HIV, hepatitis C virus (HCV), or hepatitis D virus (HDV)
* Moderate or severe renal impairment
* Recent history of pancreatitis
* Therapy with interferon, thymosin alpha or other immuno-stimulators within 24 weeks of being assigned to study drug into this study
* Prior entecavir/tenofovir combination therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2010-05; Primary Completion 2012-11 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (26):
- France (4):
  - Local Institution, Clichy
  - Local Institution, Lyon
  - Local Institution, Orléans
  - Local Institution, Strasbourg
- Germany (6):
  - Local Institution, Berlin
  - Local Institution, Hamburg
  - Local Institution, Hanover
  - Local Institution, Heindelberg
  - Local Institution, München
  - Local Institution, Tübingen
- Italy (4):
  - Local Institution, Bagno A Ripoli (Fi)
  - Local Institution, Bari
  - Local Institution, Foggia
  - Local Institution, Milan
- Netherlands (3):
  - Local Institution, Amsterdam
  - Local Institution, Arnhem
  - Local Institution, Rotterdam
- Poland (4):
  - Local Institution, Kielce
  - Local Institution, Krakow
  - Local Institution, Lodz
  - Local Institution, Wroclaw
- Romania (3):
  - Local Institution, Bucharest
  - Local Institution, Burcuresti
  - Local Institution, Timișoara
- Spain (2):
  - Local Institution, Barcelona
  - Local Institution, Valencia

REFERENCES:
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study initiated 17 May 2010; Week 48 Primary Endpoint 27 November 2012; Week 96 Study Completed18 February 2014. Participants with chronic Hepatitis B with surface antigen (HBsAg) who have been currently treated and experienced treatment failure were enrolled.
Pre-assignment Details: 144 enrolled; 92 treated. Reasons for 52 never treated: physical/laboratory test findings 30; not in target population 21; no signed consent 7; medical history/concurrent disease 2; other exclusion criteria 1; unknown 3.
Groups:
- Entecavir + Tenofovir: Entecavir (ETV) : Tablets, Oral, 1 mg, once daily, 96 weeks
  Tenofovir disoproxil fumarate (TDF): Tablets, Oral, 300 mg, once daily, 96 weeks
Period: Participants Treated With Study Drug
Arm/Group | Entecavir + Tenofovir
Started | 92
Completed | 86
Not Completed | 6
Not completed — Adverse Event | 1
Not completed — Protocol Violation | 1
Not completed — Withdrawal by Subject | 2
Not completed — Lost to Follow-up | 1
Not completed — Pregnancy | 1
Period: Post Dosing Follow-up Through 24 Weeks
Arm/Group | Entecavir + Tenofovir
Started | 85 (2 included did not complete treatment; 3 completed treatment but not included (lost to follow-up).)
Completed | 46
Not Completed | 39
Not completed — Lost to Follow-up | 1
Not completed — Withdrawal by Subject | 6
Not completed — Alternative therapy started | 32

BASELINE CHARACTERISTICS:
Population: All participants who were treated with study drug.
Groups:
- Entecavir + Tenofovir: Entecavir (ETV): Tablets, Oral, 1 mg, once daily, 96 weeks
  Tenofovir disoproxil fumarate (TDF): Tablets, Oral, 300 mg, once daily, 96 weeks
Arm/Group | Entecavir + Tenofovir
Number analyzed (Participants) | 92
Age, Continuous [Median (Full Range); unit: years] | 42.0 [18 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 69
Region of Enrollment [Number; unit: participants]
  France | 10
  Poland | 32
  Romania | 20
  Germany | 23
  Netherlands | 6
  Italy | 1
HBV DNA by PCR (log10 IU/mL) [Median (Full Range); unit: log10 IU/mL] — Hepatitis B virus deoxyribonucleic acid (HBV DNA) by polymerase chain reaction (PCR) was measured using the Roche COBAS(REGISTERED) TaqMan - High Pure System (HPS) assay. The results were reported in log 10 international units per milliliter (IU/mL), with the limit of quantification (LOQ) = 29 IU/mL and lower limit of detection (LLD) = 6 IU/mL. HBV DNA measurements were transformed by the log10 scale when analyzed as a continuous variable, using log10(LOQ-1) for values below LOQ.
  log10 IU/mL | 3.674 [1.45 to 9.30]
Baseline Hepatitis B e Antigen [Number; unit: participants]
  Positive for Hepatitis B e antigen | 56
  Negative for Hepatitis B e antigen | 34
  missing Hepatitis B e antigen test | 2
Baseline Hepatitis B e Antibody [Number; unit: participants]
  Positive for Hepatitis B e antibody | 32
  Negative for Hepatitis B e antibody | 56
  Intermediate Hepatitis B e antibody | 2
  missing Hepatitis B e antibody test | 2
Baseline Hepatitis B Surface Antigen [Number; unit: participants]
  Positive for Hepatitis B Surface Antigen | 92
  Negative for Hepatitis B Surface Antigen | 0
Baseline HBV Subtype [Number; unit: Participants]
  HBV Subtype A | 21
  HBV Subtype B | 2
  HBV Subtype C | 1
  HBV Subtype D | 35
  HBV Subtype E | 4
  HBV Subtype G | 1
  HBV Subtype H | 1
  HBV Subtype Indeterminate | 3
  Insufficient HBV DNA | 23
  Missing HBV DNA test | 1
Treatment Failure Prior to Baseline [Number; unit: participants]
  Primary Non-Response | 9
  Virological Breakthrough | 30
  Partial Virological Breakthrough | 52
  Missing | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With a Virologic Response at Week 48 - Treated Population
Description: Virologic response was defined as Hepatitis B virus (HBV) Deoxyribonucleic acid (DNA) less than 50 international units per milliliter (IU/mL); approximately 300 copies/mL. Percentage was calculated as number of participants with virologic response at Week 48 divided by the number of treated participants. Treated participants were evaluated using non-completer (NC) = failure (F). The HBV DNA by polymerase chain reaction (PCR) was measured using the Roche COBAS(REGISTERED) TaqMan - High Pure System (HPS) assay, in a central laboratory. The results were reported in IU/mL, with the limit of quantification (LOQ) = 29 IU/mL and lower limit of detection (LLD) = 6 IU/mL. HBV DNA measurements were transformed by the log10 scale when analyzed as a continuous variable, using log10(LOQ-1) for values below LOQ.
Time Frame: Week 48
Population: All treated participants were analyzed (NC = F). An exact binomial 95% confidence interval was constructed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Entecavir + Tenofovir
Number analyzed (Participants) | 92
percentage of participants | 76.1 [66.1 to 84.4]

2. Secondary Outcome: Percentage of Participants With a Virologic Response at Week 24 and at Week 96 - Treated Population
Description: Virologic response was defined as Hepatitis B virus (HBV) Deoxyribonucleic acid (DNA) less than 50 international units per milliliter (IU/mL); approximately 300 copies/mL. Percentage was calculated as number of participants with virologic response at Week 24, Week 96 divided by the number of treated participants. Treated participants were evaluated using non-completer (NC) = failure (F). The HBV DNA by polymerase chain reaction (PCR) was measured using the Roche COBAS(REGISTERED) TaqMan - High Pure System (HPS) assay. The results were reported in IU/mL, with the limit of quantification (LOQ) = 29 IU/mL and lower limit of detection (LLD) = 6 IU/mL. HBV DNA measurements were transformed by the log10 scale when analyzed as a continuous variable, using log10(LOQ-1) for values below LOQ.
Time Frame: Week 24, Week 96
Population: All treated participants were analyzed at Weeks 24 and 96 (NC = F). An exact binomial 95% confidence interval was constructed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Entecavir + Tenofovir
Number analyzed (Participants) | 92
percentage of participants
  Week 24 (n=92) | 64.1 [53.5 to 73.9]
  Week 96 (n=92) | 84.8 [75.8 to 91.4]

3. Secondary Outcome: Change From Baseline in Mean log10 HBV DNA at Weeks 12, 24, 48, and 96 - Treated Evaluable Population
Description: HBV DNA by polymerase chain reaction (PCR) was measured using the Roche COBAS(REGISTERED) TaqMan - High Pure System (HPS) assay. The results were reported in log 10 IU/mL, with the limit of quantification (LOQ) = 29 IU/mL and lower limit of detection (LLD) = 6 IU/mL. HBV DNA measurements were transformed by the log10 scale when analyzed as a continuous variable, using log10(LOQ-1) for values below LOQ. Baseline was Day 1, prior to study drug administration.
Time Frame: Baseline to Weeks 12, 24, 48, 96
Population: All treated participants with results at both baseline and on-treatment were analyzed. n=Number of treated participants with results at baseline and Week 12, Week 24, Week 48 and Week 96.
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | Entecavir + Tenofovir
Number analyzed (Participants) | 89
log10 IU/mL
  Week 12 (n=89) | -2.230 (1.5339)
  Week 24 (n=89) | -2.581 (1.8019)
  Week 48 (n=88) | -2.829 (2.0537)
  Week 96 (n=84) | -2.965 (2.1431)

4. Secondary Outcome: Percentage of Participants With HBV DNA Less Than the Lower Limit of Detection (LLD) at Weeks 24, 48, and 96 - Treated Population
Description: HBV DNA less than (<) LLD (6 IU/mL) was defined/measured by the COBAS(REGISTERED) TaqMan HPS assay at Weeks 24, 48, and 96. Percentage was calculated as number of participants with HBV DNA < LLD at Weeks 24, 48, 96 divided by the number of treated participants. Treated participants were evaluated using non-completer (NC) = failure (F).
Time Frame: Weeks 24, 48, 96
Population: All treated participants were analyzed at Weeks 24, 48 and 96 (NC = F). An exact binomial 95% confidence interval was constructed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Entecavir + Tenofovir
Number analyzed (Participants) | 92
percentage of participants
  Week 24 (n=92) | 12.0 [6.1 to 20.4]
  Week 48 (n=92) | 18.5 [11.1 to 27.9]
  Week 96 (n=92) | 16.3 [9.4 to 25.5]

5. Secondary Outcome: Percentage of Participants With Hepatitis B e Antigen (HBeAg) Loss at Weeks 24, 48, and 96 - Treated Population Who Were HBeAg Positive at Baseline
Description: Loss of HBeAg was defined as being HBeAg-negative at Weeks 24, 48, and 96 in those participants who had been HBeAg-positive at baseline. Method used for HBeAg was DiaSorin - Anti HBe enzyme immunoassay kit - procedure for qualitative determination of antibodies to HBeAg in human serum or plasma samples. Percentage was calculated as number of participants with HBeAg loss at Weeks 24 and 48 divided by the number of treated participants who were HBeAg-positive at baseline. Treated participants (HBeAg-positive at baseline) were evaluated using NC = F. Baseline was Day 1, before start of study drug.
Time Frame: Baseline to Weeks 24, 48, and 96
Population: All treated participants who were HBeAg-positive at baseline were analyzed at Weeks 24, 48 and 96 (NC = F). An exact binomial 95% confidence interval was constructed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Entecavir + Tenofovir
Number analyzed (Participants) | 56
percentage of participants
  Week 24 (n=56) | 3.6 [0.4 to 12.3]
  Week 48 (n=56) | 5.4 [1.1 to 14.9]
  Week 96 (n=56) | 8.9 [3.0 to 19.6]

6. Secondary Outcome: Percentage of Participants With HBe Seroconversion at Weeks 24, 48, and 96 - Treated Population Who Were HBeAg-positive at Baseline
Description: HBe seroconversion was defined as being both HBeAg-negative and HBeAb-positive at Weeks 24, 48, and 96 in those participants who had been HBeAg-positive at baseline. Method used was DiaSorin - Anti HBe enzyme immunoassay kit - procedure for qualitative determination of antibodies to HBeAg in human serum or plasma samples. Percentage was calculated as number of participants with HBe seroconversion at Weeks 24, 48, and 96 divided by the number of treated participants who were HBeAg-positive at baseline. Treated participants (HBeAg-positive at baseline) were evaluated using NC = F. Baseline was Day 1, before start of study drug.
Time Frame: Baseline, Weeks 24, 48, and 96
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Entecavir + Tenofovir
Number analyzed (Participants) | 56
percentage of participants
  Week 24 (n=56) | 3.6 [0.4 to 12.3]
  Week 48 (n=56) | 3.6 [0.4 to 12.3]
  Week 96 (n=56) | 1.8 [0.0 to 9.6]

7. Secondary Outcome: Percentage of Participants With Hepatitis B Surface Antigen (HBsAg) Loss at Weeks 24, 48, 96 - Treated Population Who Were HBsAg-Positive at Baseline
Description: Loss of HBsAg was defined as being HBsAg-negative at Weeks 24, 48, 96 in those participants who had been HBsAg-positive at baseline. The method used: Immunoassay - ADVIA CENTAUR from SIEMENS: in vitro diagnostic immunoassay for the qualitative and quantitative determination of HBsAg in human serum and plasma (potassium ethylene diamine tetraacetic acid, lithium or sodium heparinized). Percentage calculated as number of participants with a HBsAg loss at Weeks 24, 48, and 96 divided by the number of treated participants who were HBsAg-positive at baseline (participants were not enrolled into the study unless they were positive for HBsAg). Treated participants (HBsAg-positive at baseline) were evaluated using NC=F. Baseline was Day 1, before start of study drug.
Time Frame: Baseline, Weeks 24, 48, 96
Population: All treated participants who were HBsAg-positive at baseline and were analyzed at Weeks 24, 48, and 96 (NC = F). An exact binomial 95% Confidence Interval was constructed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Entecavir + Tenofovir
Number analyzed (Participants) | 92
percentage of participants
  Week 24 (n=92) | 1.1 [0.0 to 5.9]
  Week 48 (n=92) | 0 [NA to NA] — Confidence interval was not performed because the number of participants at Week 48 was 0.
  Week 96 (n=92) | 2.2 [0.3 to 7.6]

8. Secondary Outcome: Percentage of Participants With Hepatitis B Surface Antigen (HBsAg) Seroconversion at Weeks 24, 48, and 96 - Treated Population Who Were HBsAg-Positive at Baseline
Description: HBsAg seroconversion was defined as being both HBsAg-negative and HBsAb-positive at Weeks 24, 48, and 96 in those participants who had been HBsAg-positive at baseline. Percentage was calculated as number of participants with HBs seroconversion at Weeks 24 and 48 divided by the number of treated participants who were HBsAg-positive at baseline. Positive result for HBsAg was one of the inclusion criteria. Treated participants (HBsAg positive at baseline) were evaluated using NC=F. The method used was an Immunoassay testing - ADVIA CENTAUR from SIEMENS: in vitro diagnostic immunoassay for the qualitative and quantitative determination of HBsAg in human serum and plasma [potassium ethylenediaminetetraacetic acid (EDTA), lithium or sodium heparinized]. Baseline was Day 1, before start of study drug.
Time Frame: Baseline, Weeks 24, 48, and 96
Population: All treated participants who were HBsAg-positive at baseline and were analyzed at Weeks 24, 48 and 96 (NC = F). An exact binomial 95% confidence interval was constructed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Entecavir + Tenofovir
Number analyzed (Participants) | 92
percentage of participants
  Week 24 (n=92) | 1.1 [0.0 to 5.9]
  Week 48 (n=92) | 0 [NA to NA] — CI was not performed because the number of participants with HBsAg loss at Week 48 was 0.
  Week 96 (n=92) | 1.1 [0.0 to 5.9]

9. Secondary Outcome: Number of Participants With Treatment Emergent Serious Adverse Events (SAEs) on Treatment, and Discontinuation of Study Drug Due to Adverse Events (AE) - Treated Population
Description: AE=any new unfavorable symptom, sign, or disease or worsening of a preexisting condition that may not have a causal relationship with treatment. SAE=a medical event that at any dose results in death, persistent or significant disability/incapacity, or drug dependency/abuse; is life-threatening, an important medical event, or a congenital anomaly/birth defect; or requires or prolongs hospitalization. Treatment-related=having certain, probable, possible, or missing relationship to study drug. Grade (Gr) 1=Mild, Gr 2=Moderate, Gr 3=Severe, Gr 4=Life-threatening or disabling, Gr 5=Death. On-treatment = on Day 1 through last dose of study therapy + 5 days.
Time Frame: Day 1 to last dose of study drug plus 5 days; up to Week 96
Population: All Treated participants were analyzed.
Measure: Number; unit: participants
Arm/Group | Entecavir + Tenofovir
Number analyzed (Participants) | 92
participants
  Treatment emergent SAE | 6
  Discontinuation of treatment due to AE | 1

10. Secondary Outcome: Number of Participants With Emergence of Genotypic Resistance to Study Drugs at Weeks 48 and 96- Treated Population
Description: Testing of HBV genotype was performed at baseline for all treated patients and for participants at Weeks 48 and 96 with primary non-response or virologic breakthrough. Emergent genotypic resistance to study drugs was defined as follows: Emergent = not detected at baseline; entecavir (ETV) resistance (ETVr): participant's sample was to have rtM204V/I/S and any substitution at rtT184, rtS202, or rtM250; tenofovir (TDF) resistance (TDFr) which was based on adefovir (ADV)-mutations: participant's sample was to have rtA181T/V, rtN236T, or (rtA194T and rtM204V/I/S). Primary non-response was defined as < 1 log10 decrease in HBV DNA from baseline on treatment at or after Week 12. Virologic breakthrough was defined as ≥ 1 log10 increase in HBV DNA over nadir on treatment, either confirmed or last on-treatment followed by discontinuation of study therapy.
Time Frame: Baseline to Weeks 48, 96
Population: All treated participants who met resistance testing criteria (primary non-response or virologic breakthrough) and were tested for resistance to both study drugs were analyzed. n = number of participants analyzed at Weeks 48 and 96.
Measure: Number; unit: participants
Arm/Group | Entecavir + Tenofovir
Number analyzed (Participants) | 7
participants
  Week 48 (n=5) | 0
  Week 96 (n=7) | 0

11. Secondary Outcome: Number of Participants on Treatment With Study Drug With Laboratory Test Abnormalities Meeting Selected Criteria on Treatment - Treated Population
Description: Selected criteria presented in each category. Upper limit of normal among all laboratory ranges (ULN); Baseline (BL); alanine transaminase (ALT); milligram per deciliter (mg/dL); milliliters per minute (mL/min); greater than (>);greater than, equal to (>=); less than (<). Creatinine data presented below were confirmed, ie, at least 2 consecutive values. On-treatment = after Day 1 through last dose of study therapy + 5 days.
Time Frame: Day 1 to last dose of study drug plus 5 days; up to Week 96
Population: N=treated participants with on-treatment laboratory test results.
Measure: Number; unit: participants
Arm/Group | Entecavir + Tenofovir
Number analyzed (Participants) | 91
participants
  ALT > 2*Baseline(N=90) | 9
  ALT > 3*Baseline(N=90) | 2
  Total bilirubin >2*Baseline (N=90) | 11
  Total bilirubin >3*Baseline (N=90) | 3
  Lipase > 3*Baseline (N=90) | 4
  Creatinine increase from BL >= 20%(N=91) | 4
  Creatinine >1.5 mg/dL (N=91) | 2
  Creatinine clearance < 50 mL/min (N=91) | 1
  Phosphate < 2.0 mg/dL (N=90) | 2
  Phosphate < 2.3 mg/dL (N=90) | 8

ADVERSE EVENTS:
Time Frame: Day 1 up to 96 Weeks
Arm/Group | Entecavir + Tenofovir
Serious Adverse Events (participants affected / at risk) | 6/92
Other Adverse Events (participants affected / at risk) | 42/92
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Entecavir + Tenofovir (N=92)
Inguinal hernia (Gastrointestinal disorders) | 1
Cataract (Eye disorders) | 1
Appendicitis (Infections and infestations) | 1
Haemorrhoids (Gastrointestinal disorders) | 1
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Radius fracture (Injury, poisoning and procedural complications) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Entecavir + Tenofovir (N=92)
Bronchitis (Infections and infestations) | 6
Nasopharyngitis (Infections and infestations) | 11
Nausea (Gastrointestinal disorders) | 8
Arthralgia (Musculoskeletal and connective tissue disorders) | 7
Abdominal pain upper (Gastrointestinal disorders) | 5
Asthenia (General disorders) | 6
Dyspepsia (Gastrointestinal disorders) | 7
Diarrhoea (Gastrointestinal disorders) | 6
Dizziness (Nervous system disorders) | 5
Headache (Nervous system disorders) | 6
Fatigue (General disorders) | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.